CLINICAL TRIAL: NCT05680805
Title: Metabolic Responses of Metformin and Genetic Polymorphisms (rs628031 and rs2282143) of Solute Carrier Family 22 Member 1 Gene in Polycystic Ovary Syndrome
Brief Title: Metabolic Responses of Metformin and Genetic Polymorphisms of SLC22A1 Gene in PCOS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: University of Dhaka (Other)
Responsible Party: Principal Investigator, MA Hasanat, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2022/9559-768
Record Dates: First submitted 2022-10-27; First posted 2023-01-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome; Metformin
Keywords: Metformin; solute carrier family 22 member 1; Polycystic ovary syndrome; Metabolic response
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCOS (Experimental): Participants with PCOS
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin 1500 mg/day in 3 divided dose for 24 weeks

SUMMARY:
The aim of this study is to see the associations of metabolic responses of metformin with single nucleotide polymorphisms (SNPs) (rs628031 and rs2282143) of solute carrier family 22 member 1 (SLC22A1) gene in women with polycystic ovary syndrome (PCOS). This prospective clinical study will be conducted in the department of Endocrinology, Bangabandhu Sheikh Mujib Medical University (BSMMU) from February 2023 to September 2024 over a period of two years. A total of at least 100 women with PCOS (18 - 35 years) diagnosed based on International Evidence-based Guideline for PCOS 2018, will be included consecutively by convenient sampling. After taking informed written consent, relevant clinical history will be taken and physical examinations will be done at baseline. Following a run in phase of three weeks, patients will visit thrice after 1, 12 & 24 weeks of metformin maintenance therapy with a window period of 14 days both ways. Blood samples will be collected in fasting state at baseline and after 24 weeks of treatment to measure glycemic status, lipid profile, fasting insulin, c-peptide and detection of SLC22A1 gene (rs628031 and rs2282143) polymorphisms. Glucose will be measured by glucose oxidase method, lipids by glycerol phosphate dehydrogenase peroxidase method, insulin by chemiluminescent microparticle immunoassay, c-peptide by enzyme-linked immunosorbent assay (ELISA) and genetic analysis of rs628031 and rs2282143 by polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP).

DETAILED DESCRIPTION:
Objectives of the Study General objective Determination of the association of metabolic responses to metformin with SLC22A1 gene polymorphisms (rs628031 and rs2282143) in women with PCOS Specific objectives

* To see the changes of metabolic profile (body mass index, waist circumference, blood pressure, glycemic status, insulin resistance, c-peptide and lipid) in 24 weeks of metformin therapy in women with PCOS
* Determination of frequency of SLC22A1 gene polymorphisms (rs628031 and rs2282143) in women with PCOS
* Categorization of PCOS patients according to SLC22A1 gene polymorphisms (rs628031 and rs2282143) into wild and variant groups
* Comparison of metabolic changes of 24 weeks of metformin therapy between wild vs. variant group of SLC22A1 gene polymorphisms (rs628031 and rs2282143) in women with PCOS

Others:

* Determination of the short-term side-effects of metformin in women with PCOS
* Comparison of metformin side-effects in women with PCOS with or without SLC22A1 gene polymorphisms (rs628031 and rs2282143)

Materials and Methods:

Type of study:

Prospective clinical study

Place of study:

Department of Endocrinology, BSMMU

Study period:

October 2022 to September 2024

Study population:

Reproductive aged (18 - 35 years) women of PCOS

Sampling method:

Consecutive purposive/convenient sampling

Sample size:

The sample size will be calculated from following formula:

n= {(Zα + Zβ)^2 × (σ1^2 + σ2^2)} ÷ (μ1 - μ2)^2 From a previous similar study, the 2 hours OGTT glucose/insulin ratio (GIR) before and after 24 weeks of metformin therapy were 2.3±2.5 and 3.2±3.2 in variant genotype and 2.0±1.9 and 3.9±2.9 respectively in wild genotype of SLC22A1 rs628031. The mean differences in variant and wild genotype were 0.9±0.7 and 1.9±1.0 respectively.

Here, Zα= 1.96 at 95% confidence level, Zβ= 1.28 at 90% power, μ1= mean changes of GIR after metformin in variant genotype of rs628031 (AG/GG) = 0.9, μ2 = mean of GIR after metformin in wild genotype of rs628031(AA) = 1.9, Assuming standard deviation (SD)= 1.5 (σ1=σ2) in both groups

Minimum number of sample to be studied in each group, n= {(1.96 + 1.28)^2 × (1.52 + 1.52)} ÷ (0.9 - 1.9)^2

* {(3.24)^2 × (2.25 + 2.25)} ÷ (1.0)^2
* {10.50 × 4.50} ÷ 1 = 47.25 ÷ 1 = 47.25 At least 94 patients with PCOS are required for this study. However considering dropout, at least 100 patients with PCOS will be taken for the study. Sample size may be increased if required.

Study procedure Newly diagnosed at least 100 women of reproductive age (18 - 35 years) PCOS patients will be consecutively recruited from the department of Endocrinology, BSMMU. Informed written consent will be taken from patients and asked to come in fasting state on particular day, time and place twice a week. Related history (reproductive, personal and family history) will be taken and physical examination (height, weight, waist circumference, hip circumference, acne, hirsutism, acanthosis nigricans) will be done and all data will be documented in a pretested semi-structured questionnaire.

Blood sample collection at baseline:

About 10 ml of venous blood will be drawn from each participant with 8 - 12 hours of fasting. Then a 75 gm oral glucose tolerance test (OGTT) will be done and another five ml of blood will be collected after two hours. About two ml of blood collected during fasting and two hours after OGTT will be kept in fluorinated tube for blood glucose measurement on the same day of collection. Additional two ml of whole blood will be preserved at -70 degree Celcius in the department of Endocrinology for polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP) after completing all biochemical analysis to avoid bias. Remaining six ml blood collected during fasting and three ml of blood collected after OGTT will be kept standing for 15 minutes to allow clotting. After centrifugation, serum will be separated and kept into eppendorf. After proper labeling, they will be preserved in a -700C refrigerator. Biochemical analysis (glucose and lipid profile) of the serum will be done on the same day and insulin and c-peptide within seven days of collection.

Interventions Lifestyle modifications Patients will be counseled at the time of diagnosis and a written document will be provided.

Diet

* An individualized diet chart prepared by dietitian will be provided
* Overweight/obese: An energy deficit of 500 Kcal/day diet from weight maintenance diet
* Others: Weight maintenance diet Physical activity
* A minimum of 150 minutes/week of moderate intensity physical activity (brisk walking at a rate of 6 km/h) with muscle strengthening activities on 2 non-consecutive days/week
* activity be performed in at least 10-minute bouts or around 1000 steps, aiming to achieve at least 30 minutes daily at least 5 days a week

Metformin prescription Ingredients of each tablet of metformin Each tablet of metformin contains metformin 500 mg HCl, BP along with inactive ingredients of povidone, microcrystalline cellulose, croscarmellose sodium and magnesium stearate. In addition, the coating for the tablets contains polyethylene glycol, polyvinyl alcohol, titanium dioxide, talc, gum acacia, maltodextrin, propylene glycol and natural flavors.

Inventory All the tablets of metformin will be dispensed periodically to the study participants by the researcher at baseline and 1st visit (after week 1) and 2nd follow up visit after 12 weeks of metformin maintenance therapy (1500 mg/day). Metformin tablets will be preserved as per the instructions of manufacturer. Expiry date and quality of the drugs will be checked periodically.

Run-in phase Metformin will be prescribed at 500 mg once daily after dinner and will increase to 1500 mg/day in three divided doses after main meals within two weeks of initiation. Patients will be asked to come with a chart of drug compliance and side-effects one week after initiation of 1500 mg/day of metformin. Patients who will not able to tolerate 1500 mg/day, be excluded from the study for analysis of metabolic responses.

Maintenance dose: 1500 mg/day in three divided dose for 24 weeks Follow up: Patients will be requested to come for three follow up visits after 1, 12 and 24 weeks of maintenance metformin therapy with a window period of two weeks both ways. During 1st follow up visit (after 1 week) patients' drug compliance and side-effects will be monitored; clinical status along with lifestyle and drug's compliance and adverse effects will be documented after 12 weeks (2nd follow up visit). After 24 weeks (3rd visit), patient's biochemical metabolic profiles will also be done with above mentioned clinical information.

Blood sample collection after 24 weeks About eight ml of venous blood after 24 weeks of metformin therapy with 8 - 12 hours of fasting will be collected to measure FBG, HbA1C, insulin, c-peptide and lipid profile and a 75 gm OGTT followed by five ml of blood will be collected for measurement of glucose and insulin.

Drug compliance:

It will be monitored over phone weekly for the first two weeks and then each visit to the researcher. Patients will be requested to come with empty blisters of metformin. A record book will be maintained to monitor compliance properly. Patients with drug compliance <95% at any time of the study will be excluded from the analysis for metabolic responses.

Adverse events monitoring:

On each visit patients will be provided with an adverse event (AE) diary for noting pre-specified gastro-intestinal (GI) events. They will also be asked for any serious adverse effect (SAE) or other AE apart from GI event. All AE and SAE will be recorded in given AE form and will be preserved in patients' files. Patients will be advised to strictly use barrier contraception. Serum ALT and creatinine will be measured after 24 weeks of metformin therapy also.

ELIGIBILITY:
Inclusion Criteria:

* • Newly diagnosed women of reproductive age (18 - 35 years) PCOS patients

Exclusion Criteria:

* • Patients having known similar endocrine disorders (hypothyroidism, hyperprolactinemia, androgen producing tumor, congenital adrenal hyperplasia, etc)

  * Planning to conceive within next six months, pregnant/ lactating mother
  * Patients with known diabetes mellitus, ischemic heart disease, chronic liver (serum ALT >2 × upper limit of normal) and renal disease (eGFR <60 ml/minute/1.73 m2 body surface area)
  * Patients taking oral contraceptive, steroid or drugs affecting insulin resistance (metformin, pioglitazone)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin resistance (HOMA-IR) | 24 weeks
  Insulin resistance
Lipid profile | 24 weeks
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglyceride, all in mg/dL
Weight | 24 weeks
  Weight (Kg)
C-peptide | 24 weeks
  Beta cell secretory capacity, ng/ml
SLC22A1 (rs628031) | 24 weeks
  AA, AT, TT- frequency
SLC22A1 (rs2282143) | 24 weeks
  CC, CG, GG- frequency
Glycemic status | 24 weeks
  Fasting plasma glucose (mmol/L), 2 hours after OGTT (2H-OGTT) glucose (mmol/L)
Height | 24 weeks
  Height (meter)
Waist circumference | 24 weeks
  waist circumference (cm)
Systolic blood pressure | 24 weeks
  Systolic blood pressure (mm-Hg)
Diastolic blood pressure | 24 weeks
  Diastolic blood pressure (mm-Hg)

SECONDARY OUTCOMES:
Number of participants with side-effects | 24 weeks
  Number of participants with nausea, vomiting, diarrhea, loose motion, and others

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Hasanat, MPhil, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Department of Endocrinology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Only group data

REFERENCES:
- [Result] Gambineri A, Tomassoni F, Gasparini DI, Di Rocco A, Mantovani V, Pagotto U, Altieri P, Sanna S, Fulghesu AM, Pasquali R. Organic cation transporter 1 polymorphisms predict the metabolic response to metformin in women with the polycystic ovary syndrome. J Clin Endocrinol Metab. 2010 Oct;95(10):E204-8. doi: 10.1210/jc.2010-0145. Epub 2010 Jul 21. PMID 20660041
- [Result] Chang HH, Hsueh YS, Cheng YW, Ou HT, Wu MH. Association between Polymorphisms of OCT1 and Metabolic Response to Metformin in Women with Polycystic Ovary Syndrome. Int J Mol Sci. 2019 Apr 7;20(7):1720. doi: 10.3390/ijms20071720. PMID 30959948
- [Result] Schweighofer N, Lerchbaum E, Trummer O, Schwetz V, Pieber T, Obermayer-Pietsch B. Metformin resistance alleles in polycystic ovary syndrome: pattern and association with glucose metabolism. Pharmacogenomics. 2014 Feb;15(3):305-17. doi: 10.2217/pgs.13.223. PMID 24533710